CLINICAL TRIAL: NCT03023631
Title: Human Papillomavirus Antibody Response After GARDASIL 9 Vaccination in Patients After Allogeneic Stem Cell Transplantation
Brief Title: Gardasil 9 Vaccine in Preventing HPV Infection in Patients With Hematologic Malignancies Undergoing Donor Stem Cell Transplant
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0714; NCI-2018-02606 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0714 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-13; First posted 2017-01-18 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplant Recipient; Hematopoietic and Lymphoid Cell Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prevention (Gardasil 9 vaccine) (Experimental): Patients undergo standard of care allogeneic stem cell transplant. 6-12 months following transplant, patients receive recombinant human papillomavirus nonavalent vaccine IM on day 0 and at 2 and 6 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Recombinant Human Papillomavirus Nonavalent Vaccine

INTERVENTIONS:
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV VLP Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine

SUMMARY:
This phase IV trial studies how well Gardasil 9 vaccine works in preventing human papillomavirus (HPV) infection in patients with hematologic malignancies who are undergoing donor stem cell transplant. Vaccines, such as Gardasil 9, may help the body build an effective immune response to kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the immunogenicity of recombinant human papillomavirus nonavalent vaccine (GARDASIL 9) administered after allogeneic stem cell transplant (SCT) in patients with hematologic malignancy by comparing HPV 9-plex competitive Luminex immunoassay (9-plex cLIA) titers before and after GARDASIL 9 administration.

II. To evaluate the safety and tolerability of GARDASIL 9 administered after allogeneic SCT in patients with hematologic malignancy.

OUTLINE:

Patients undergo standard of care allogeneic stem cell transplant. 6-12 months following transplant, patients receive recombinant human papillomavirus nonavalent vaccine intramuscularly (IM) on day 0 and at 2 and 6 months in the absence of disease progression or unacceptable toxicity.

After completion of study intervention, patients are followed up within 3 days.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking adult MD Anderson patients with hematologic malignancy at 6-12 months +/- 8 weeks post allogeneic stem cell transplantation who will receive usual post-stem cell transplant vaccinations
* All patients from approved protocol 2015-0795 will be invited to this vaccine study

Exclusion Criteria:

* Prior allogeneic SCT
* Platelet count less than or equal to 25,000 K/uL
* Absolute neutrophil count less than or equal to 500/uL
* Patients who have ever received HPV vaccination (at least one dose of HPV vaccine)
* Patients with a prior history of HPV-related malignancy
* Female patients who tested positive for pregnancy during pre-SCT evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Antibody response defined as numerically elevated antibody titer of any type at 1 month post-dose 3 (month 7) | At 1 month post-dose 3
  Antibody response at 1 month post-dose 3 (month 7) will be compared with baseline antibody level. The study will use results from the 9-plex competitive Luminex immunoassay (9-plex cLIA) test to estimate the antibody response rate at dose 3 with 95% confidence interval (CI). Will apply Student t-test/Wilcoxon test to compare continuous variables between patients who obtained antibody response as defined in the primary endpoint (responders) and those who did not respond (non-responders), and the chi-square test or the Fisher's exact test to assess the association between response status and patients' demographic and clinical characteristics. Logistic regression analysis will be used to assess the multivariate relationship between patient demographic and clinical characteristics on the probability of antibody response.

SECONDARY OUTCOMES:
Incidence of adverse events graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 | Up to 3 days post-intervention
  Safety and tolerability of recombinant human papillomavirus nonavalent vaccine measured by occurrence of grade >= 3 adverse events (AEs) that are possibly, probably, or definitely related to recombinant human papillomavirus nonavalent vaccine for all 3 vaccine administrations. The study will report the AE rate with a corresponding upper bound of a 1-sided 95% CI.
Antibody persistence at 6 months post-dose 3 | At 6 months post-dose 3
  Antibody persistence at 6 months post-dose 3 will be compared with 1 month post-dose 3. The study will apply a paired t-test with noninferiority hypotheses.
Human papillomavirus (HPV) vaccination completion rate | Up to 3 days post-intervention
  The study will calculate the proportion of patients who are able to complete the 3 shot series of HPV vaccination. Will describe them in terms of demographics, and clinical characteristics.
Estimation of antibody titers | At 6-12 months post-transplant, and at 1 and 6 months post-dose 3
  Antibody titer will be measured repeatedly by the 9-plex cLIA test. Appropriate transformation (e.g. log transformation) of antibody titer will be used in the analyses to satisfy the normality assumption of linear or linear mixed effect model. Geometric mean titers will be used to summarize antibody titer at each time point. Linear mixed effect models for repeated measures analysis will be employed to assess change in antibody titer over time and to compare antibody titer change over time between different patient groups adjusting for other important covariates including disease characteristics (tumor stage, site, pathology), and other patient prognostic factors. Interaction between time and patients' characteristics on the change of antibody titer will be also investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica P Hwang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org